CLINICAL TRIAL: NCT06710262
Title: T-TAS® wS Method Comparison
Status: Completed | Type: Observational
Sponsor: Hikari Dx, Inc. (Other)
Collaborators: ZACROS Corporation (Unknown)
Responsible Party: Sponsor
Other Study IDs: NX-VAP-AP-I0001
Record Dates: First submitted 2024-11-20; First posted 2024-11-29 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Antiplatelet Therapy; Healthy Donors; Von Willebrand Disease (VWD)
Keywords: T-TAS; Primary hemostasis
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Healthy donors: Subjects with no evidence of primary hemostasis abnormalities
  Interventions: Diagnostic Test: T-TAS PL Assay
- Aspirin monotherapy: Subjects taking aspirin monotherapy
  Interventions: Diagnostic Test: T-TAS PL Assay
- Dual antiplatelet therapy: Subjects taking dual antiplatelet therapy (aspirin plus either clopidogrel, prasugrel, or ticagrelor)
  Interventions: Diagnostic Test: T-TAS PL Assay
- Von Willebrand Disease: Subjects with a prior diagnosis of Von Willebrand Disease
  Interventions: Diagnostic Test: T-TAS PL Assay

INTERVENTIONS:
Diagnostic Test: T-TAS PL Assay — The T-TAS PL assay is a flow chamber assay for measuring primary hemostatic function

SUMMARY:
This study involves the collection of blood samples and measurement with the T-TAS PL assay to compare the performance of the T-TAS wS instrument to the T-TAS 01 instrument

DETAILED DESCRIPTION:
This study will compare PL assay measurements obtained with the T-TAS wS instrument (subject device) with PL assay measurements obtained with the T-TAS 01 instrument (predicate method). The T-TAS PL assay will be used to facilitate the comparison between instruments using intended use blood samples from the intended use population. The study will be conducted at a minimum of 3 locations in the United States and will enroll up to 120 subjects. The following subject populations will be enrolled into the study (minimum enrollment numbers indicated in parentheses):

* Ostensibly healthy subjects
* Subjects taking 81 mg or higher daily aspirin monotherapy (ASA)
* Subjects taking dual antiplatelet therapy (DAPT)
* Subjects with von Willebrand disease (VWD)

ELIGIBILITY:
Ostensibly Healthy Donors

Inclusion Criteria:

* Males and females age 21 years or older.
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Hospitalization or doctor's visits within prior 30 days, except for routine checkup/physical examination.
* Use of antiplatelet therapy within the past 7 days, e.g. aspirin, clopidogrel, prasugrel, ticagrelor, cilostazol.
* Use of anticoagulant drugs within the past 7 days, e.g. heparin, bivalirudin, warfarin, rivaroxaban, and apixaban.
* Use of certain nonsteroidal anti-inflammatory drugs (NSAIDs) that inhibit COX-1 such as naproxen or ibuprofen within the past 3 days, unless confirmed to not inhibit platelet activity (such as celecoxib).
* History of anemia.
* Known thrombocytopenia (platelet count < 100,000/μL).
* Significant renal dysfunction or dialysis.
* History of platelet disorders e.g. von Willebrand factor deficiency, Glanzmann's thrombasthenia or Bernard-Soulier syndrome.
* History of hemophilia or bleeding disorders.
* Known active gastrointestinal disease including peptic ulcers, gastro-esophageal reflux disease (GERD), and hyperacidity.
* Currently participating in a study involving an investigational drug or compound known to affect coagulation or hemostasis.
* Subjects with significant past medical history as determined by the Investigator that would pose safety concerns or interfere with the study goals.

Antiplatelet Therapy Subjects

Inclusion Criteria:

* Males and females age 21 years or older.
* One of the following antiplatelet therapy regimens:
* Aspirin monotherapy:
* 81 mg or higher aspirin daily for 1 or more days
* Dual antiplatelet therapy:
* 81 mg or higher aspirin plus either 1) ≥300 mg clopidogrel loading dose within the prior 5 days followed by 75 mg daily clopidogrel, or 2) 75 mg daily clopidogrel daily for ≥5 days.
* 81 mg or higher aspirin plus either 1) 60 mg prasugrel loading dose within the prior 5 days followed by either 5 or 10 mg daily prasugrel, or 2) 5 or 10 mg daily prasugrel daily for ≥5 days.
* 81 mg aspirin plus either 1) 180 mg ticagrelor loading dose within the prior 5 days followed by 2x90 mg daily ticagrelor, or 2) 2x90 mg daily ticagrelor daily for ≥5 days.
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Use of antiplatelet therapy other than aspirin, clopidogrel, prasugrel, or ticagrelor (e.g. cilostazol, abciximab, eptifibatide) within the past 7 days.
* Use of anticoagulant drugs within the past 7 days, e.g. heparin, bivalirudin, warfarin, rivaroxaban, and apixaban.
* Significant renal dysfunction or dialysis.
* Known thrombocytopenia (platelet count < 100,000/μL).
* History of platelet disorders e.g. von Willebrand factor deficiency, Glanzmann thrombasthenia or Bernard-Soulier syndrome.
* History of hemophilia or bleeding disorders.
* Females who are in the last trimester of pregnancy or are breastfeeding.
* Known active gastrointestinal disease including peptic ulcers, gastro-esophageal reflux disease (GERD), and hyperacidity.
* Currently participating in a study involving an investigational drug or compound known to affect coagulation or hemostasis.
* Subjects with significant past medical history as determined by the Investigator that would pose safety concerns or interfere with the study goals.

Von Willebrand Disease Subjects

Inclusion Criteria:

* Males and females age 21 years or older.
* Prior diagnosis of von Willebrand disease type 1, 2A, 2B, 2M, or 3
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Prior diagnosis of von Willebrand disease type 2N
* Use of antiplatelet therapy besides aspirin within the past 14 days.
* Use of anticoagulant drugs within the past 14 days, e.g. heparin, bivalirudin, warfarin, rivaroxaban, and apixaban.
* Use of certain nonsteroidal anti-inflammatory drugs (NSAIDs) that inhibit COX-1 such as naproxen or ibuprofen within the past 7 days, unless confirmed to not inhibit platelet activity (such as celecoxib).
* Significant renal dysfunction or dialysis.
* Known thrombocytopenia (platelet count < 100,000/μL).
* Currently participating in a study involving an investigational drug or compound known to affect coagulation or hemostasis.
* Subjects with significant past medical history as determined by the Investigator that would pose safety concerns or interfere with the study goals.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital or clinic patients, healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2024-08-21 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Method agreement | For each enrolled subject, following testing of blood sample with the T-TAS PL assay; data will be compiled and analyzed in aggregate at the time of study completion.
  Agreement of PL assay AUC results between the T-TAS wS and T-TAS 01 measurement systems

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Florida Health Jacksonville, Jacksonville, Florida
  - Sinai Hospital of Baltimore, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No
Results may be proprietary and/or used to support regulatory submissions